CLINICAL TRIAL: NCT02493998
Title: A Prospective, Observational Study of Mucopolysaccharidosis Type IIIB (MPS IIIB)
Brief Title: A Study of Mucopolysaccharidosis Type IIIB (MPS IIIB)
Status: Completed | Type: Observational
Sponsor: Allievex Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 250-901
Record Dates: First submitted 2015-06-22; First posted 2015-07-10 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Mucopolysaccharidosis Type IIIB; Mucopolysaccharidosis Type 3 B; MPS III B; MPS 3 B
Keywords: Sanfilippo Syndrome Type B
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mucopolysaccharidosis type IIIB (MPS IIIB, also known as Sanfilippo Syndrome Type B) is a severe neurodegenerative disorder. The purpose of this study is to learn more about the health problems in patients with MPS IIIB and how to measure these problems over time. It will particularly look at how the disease develops in young children. This is an observational study, so no experimental drug will be given. The results from this study will help us design future studies to measure whether these health problems get better when we give experimental drug for MPS IIIB.

DETAILED DESCRIPTION:
This is a multicenter, multinational, longitudinal, observational study in subjects 1 through 10 years of age who have been diagnosed with MPS IIIB. Data will be prospectively collected from 20 to 30 subjects to understand the clinical progression of MPS IIIB in terms of neurocognitive function, behavior, quality of life, imaging characteristics, genotype, and biochemical markers of disease burden. This information may help inform the design and interpretation of subsequent interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Individuals eligible to participate in this study must meet all of the following criteria:
* Has deficient NAGLU enzyme activity at Screening. Blood for NAGLU enzyme activity will be collected and analyzed centrally.
* Is ≥ 1 and ≤ 10 years of age and has an age-equivalent of ≥ 12 months on the VABS-II
* DQ ≥ 50 (determined by BSID-III or KABC-II)
* Has presented with signs/symptoms consistent with MPS IIIB; for individuals who have not presented with signs/symptoms of disease (e.g., siblings of known patients), the determination of eligibility will be at the discretion of the BioMarin medical monitor in conjunction with the site investigator.
* Written informed consent from parent or legal guardian and assent from subject, if required
* Has the ability to comply with protocol requirements, in the opinion of the investigator

Exclusion Criteria:

* Has another neurological illness that may have caused cognitive decline (e.g., trauma, meningitis, or hemorrhage) before study entry
* Requires ventilation support, except for noninvasive support at night
* Has received stem cell, gene therapy or ERT for MPS IIIB
* Has contraindications for neurosurgery (e.g., congenital heart disease, severe respiratory impairment, or clotting abnormalities)
* Has contraindications for MRI scans (e.g., cardiac pacemaker, metal fragment or chip in the eye, or aneurysm clip in the brain)
* Has a history of poorly controlled seizure disorder
* Is prone to complications from intraventricular drug administration, including patients with hydrocephalus or ventricular shunts
* Has received any investigational medication within 30 days prior to the Baseline visit or is scheduled to receive any investigational drug during the course of the study
* Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with protocol requirements, the subject's wellbeing or safety, or the interpretability of the subject's clinical data.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study Population: Subjects diagnosed with MPS IIIB
  Males and females 1 through 10 years of age (ie, until they turn 11) with a documented diagnosis of MPS IIIB are eligible to participate in this observational study. Up to approximately 5 subjects 6 to 10 years old, inclusive, will be enrolled; the remaining subjects will be 1 to 5 years old, inclusive. Additional entry criteria follow.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Neurocognitive function | Screening, baseline, and every 12 weeks, for up to 48-96 weeks
  A neurodevelopmental assessment will be performed using standardized developmental tests to provide quantifiable measures of neurocognitive function.
Imaging characteristics | Baseline and every 24 weeks, for up to 48-96 weeks
  MRI will be used to assess changes in size of various organs affected by the disease, including brain, liver and spleen.
Behavioral function | Baseline and every 12 weeks, for up to 48-96 weeks
  Disease-related behaviors will be assessed using an MPS III-specific behavior rating scale.
Hearing | Baseline and every 24 weeks, for up to 48-96 weeks
  The function of conductive and sensorineural hearing pathways will be assessed using tympanometry and auditory brainstem response (ABR).
Sleep habits | Baseline and every 24 weeks, for up to 48-96 weeks
  Patient sleep habits will be assessed using specific questionnaires.
Quality-of-life | Baseline and every 24 weeks, for up to 48-96 weeks
  Multiple QOL tools will be used to capture physical, mental, and social well-being of the patient as well as to examine the impact of the patient's disease on the parent/guardian and family.
Biochemical, Molecular, Cellular and Genetic Markers of Disease Burden | Baseline and every 24 weeks, for up to 48-96 weeks
  Blood, urine, and CSF samples will be used to evaluate biochemical, molecular cellular, and genetic/genomic aspects of MPS IIIB.

CONTACTS AND LOCATIONS:
Overall Officials: Allievex Medical Monitor, Study Director — Allievex Corporation
Locations (8):
- Children's Hospital and Research Center Oakland, Oakland, California, United States
- Melbourne Children's Trials Centre, Melbourne, Victoria, Australia
- Fundacion Cardioinfantil-Instituto de Cardiologia, Bogotá, Colombia
- University Medical Center Hamburg Eppendorf, Department of Pediatrics, Hamburg, Germany
- Hospital Clinico Universitario de Santiago, Santiago de Compostela, Spain
- MacKay Memorial Children's Hospital, Taipei, Taiwan
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)
- Somers Clinical Research Facility, Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Derived] Okur I, Ezgu F, Giugliani R, Muschol N, Koehn A, Amartino H, Harmatz P, de Castro Lopez MJ, Couce ML, Lin SP, Batzios S, Cleary M, Solano M, Peters H, Lee J, Nestrasil I, Shaywitz AJ, Maricich SM, Kuca B, Kovalchin J, Zanelli E. Longitudinal Natural History of Pediatric Subjects Affected with Mucopolysaccharidosis IIIB. J Pediatr. 2022 Oct;249:50-58.e2. doi: 10.1016/j.jpeds.2022.06.005. Epub 2022 Jun 13. PMID 35709957